CLINICAL TRIAL: NCT04149366
Title: Clinical and Radiographic Evaluation of Different Thickness of Vacuum Formed Retainer (Essix Retainer) During Retention Phase After Orthodontic Treatment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mostafa Ahmed, assistant lecturer, Minia University
Other Study IDs: 295
Record Dates: First submitted 2019-10-27; First posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Temporomandibular Joint Disorders After Using Essix Retainer
MeSH Terms: interventions — Orthodontic Retainers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- group 1 (Wrapround retainer)
  Interventions: Device: Retainer
- Group 2 (Essix retainer 1mm)
- Group 3 (Essix retainer 1.5 mm)
- Group 3 (Essix retainer 2mm)

INTERVENTIONS:
Device: Retainer — Orthodontic retainer
  Groups: group 1 (Wrapround retainer)

SUMMARY:
vacuum formed retainer act as bite raiser that increase vertical dimension which may affect Tempromandibular joint and aim of this study is to perform clinical and radiographic evaluation of different thickness of vacuum formed retainer (Essix retainer) during retention phase after orthodontic treatment

ELIGIBILITY:
Inclusion Criteria:

* patients finished fixed orthodontic treatment with no signs or symptoms of temporomandibular joint disorders
* patients indicated for removable retainer

Exclusion Criteria:

* any systemic disease
* chronic medication uptake
* bad oral hygiene pathological conditions of temporomandibular joint

Ages: 15 Years to 35 Years | Sex: All
Age Groups: Child, Adult
Study Population: patients that have finished fixed orthodontic treatment with no signs or symptoms of temporomandibular joint disorders
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-10-29 (Estimated); Primary Completion 2020-08-25 (Estimated); Study Completion 2020-10-25 (Estimated)

PRIMARY OUTCOMES:
Clinical effect of retainer on temporomandibular joint | 9 months
  Absence of pain, deviation and trismus
Radiographic effect of retainer on tempromandibular joint | 9 months
  Normal dissc position